# **ABBOTT**

#### **Statistical Analysis Plan**

# Module 1 (Non-standard data and analyses)

Version 3.0, Date 19Sep2017

Study: DYDR3004 (formerly M13-625)

A Randomized, Open-label, Two-arm, Multicenter Study Comparing the Efficacy, Safety and Tolerability of Oral Dydrogesterone 30 mg daily versus Crinone 8% intravaginal progesterone gel 90 mg daily for Luteal Support in In-Vitro Fertilization (LOTUS II)





## TABLE OF CONTENTS

| SIGNA | TURE PAGE | 2 |
|-------|-----------------------------------------------------------|----|
| 1. | ABBREVIATIONS | 7 |
| 1.1 | Standard Abbreviations | |
| 2. | INTRODUCTION | 9 |
| 3. | SUMMARY OF THE PROTOCOL | 10 |
| 3.1 | Overall Study Plan | |
| 3.2 | Study Flowchart | |
| 3.3 | Study Objectives | 11 |
| 3.4 | Sample Size and Randomization | |
| 4. | STATISTICAL ANALYSIS | 13 |
| 4.1 | Subject samples | 13 |
| 4.2 | Efficacy analysis | |
| 4.2.1 | Calculation of Pregnancy Rates | |
| 4.2.2 | Primary Efficacy Analysis | |
| 4.2.3 | Secondary efficacy analysis | |
| 4.2.4 | Other efficacy analysis | |
| 4.3 | Safety analysis | |
| 4.4 | Interim Analysis | |
| 4.5 | Data Safety Monitoring Board | |
| 4.6 | Safety Management Team | |
| 5. | DESCRIPTION OF NON-STANDARD DATA COLLECTED AND | |
| | DERIVED VARIABLES | |
| 5.1 | Other Non-Standard Baseline Characteristics | |
| 5.2 | Non-Standard Disease History | |
| 5.3 | Efficacy data | |
| 5.4 | Non-standard Safety Data | 24 |
| 5.5 | Drug Accountability and Exposure | |
| 5.5.1 | Drug Accountability | |
| 5.5.2 | Exposure | 24 |
| 6. | FURTHER SPECIFICATIONS TO THE STANDARD ANALYSES IN | |
| | MODULE 2 | |
| 6.1 | Trial Design [2] | |
| 6.1.1 | Trial Periods | |
| 6.1.2 | Trial Elements | |
| 6.1.3 | Trial Arms | |
| 6.1.4 | Unique Treatments | |
| 6.1.5 | Visits and related definitions | |
| 6.2 | Further Specifications to the Standard Tables in Module 2 | |
| 6.3 | Other Further Specifications | 29 |

| 7. | CHANGES TO PLANNED ANALYSES | |
|---------------|------------------------------------------------------|----|
| 7.1 | Changes to the Analysis as Laid Down in the Protocol | |
| 7.2 | Changes from SAP Version 2.0 to Version 3.0 | 30 |
| 8. | REFERENCE | 31 |
| 0 | A DDENIDICES | 22 |
| <b>9.</b> 9.1 | APPENDICESStudy Flowchart | |
| 9.2 | Tables, Listings and Figures | |
| 9.2.1 | Tables | 35 |
| 9.2.2 | Listings | |
| 9.2.3 | Figures | 48 |



SAP Template Version 3.0



#### 1. ABBREVIATIONS

#### 1.1 Standard Abbreviations

AE adverse event

ALAT alanine aminotransferase ASAT aspartate aminotransferase

APGAR Appearance, Pulse, Grimace, Activity, Respiration

BMI body mass index bpm beats per minute CRF case report form

CRO contract research organization
DBP diastolic blood pressure

ET embryo transfer

eCRF Electronic case retrieval form

FA Full Analysis

HCG human chorionic gonadotropin HLGT High Level Group Term

HLT High Level Term

ICH International Conference on Harmonization

IVF in vitro fertilization

IWRS/IRT interactive web response system

LDA day number of the last day of drug administration

LH luteinizing hormone LLT Lowest Level Term

max maximum

MedDRA Medical Dictionary for Regulatory Activities

min minimum

N,n number of observations

NA not applicable
PP Per Protocol
PRL Prolactin
PT Preferred Term

RBC red blood cells
SAE serious adverse event
SAP statistical analysis plan
SBP systolic blood pressure
SD standard deviation

SOC System Organ Class
SOP standard operating procedure

T Testosterone

TEAE treatment-emergent adverse event

TESAE treatment-emergent serious adverse event

tid three times daily

TLF/T,L,F tables, listings and figures TSH thyroid-stimulating hormone

WBC white blood cells

WHO-DD(E) World Health Organization – Drug Dictionary (enhanced)



#### 3. SUMMARY OF THE PROTOCOL

#### 3.1 Overall Study Plan

This is a prospective, open label, randomized, two-arm, multicenter study comparing the efficacy, safety and tolerability of the oral dydrogesterone treatment regimen versus an intravaginal micronized progesterone gel treatment for the luteal support in in-vitro fertilization (IVF).

The study will be conducted according to the following scheme:

- Visit 1 (Day -40 to -1 (according to amendment 2)/or Day -14 to -1 if the study is conducted according to amendment 1[day of downregulation/ovarian follicle stimulation]): Screening and Enrollment

Subjects signing the informed consent form will be evaluated for eligibility. They will undergo a physical examination including vital signs; a review of their medical history and concomitant medication. A transvaginal ultrasound will be done, if the last transvaginal examination is older than 14 days. Blood samples will be taken for baseline routine laboratory values. For patients conducting the study according to amendment 3 hormone testing should also be performed for subjects where FSH, estradiol ( $E_{2}$ ), LH (luteinizing hormone), PRL (Prolactin), T (Testosterone) and TSH (thyroid-stimulating hormone) are not available prior screening.

- Treatment period (Day 1 to Week 10):

Luteal support starts on Day 1 (Visit 2), the day of oocyte retrieval. Subjects will be treated with one of the following treatment regimens:

#### Group I

Oral Dydrogesterone 10 mg tablets three times daily (tid) (Duphaston) or

#### **Group II**

Crinone 8%, intravaginal progesterone gel 90 mg, once daily

- Visit 3 (Day 3 - 6): Day of embryo transfer

This interventional treatment is following the clinic specific in vitro fertilization (IVF) protocol.

- Visit 4 (Day 17 – 20 (according to amendment 2)/or Day 15 +/- 3 days if the study is conducted according to amendment 1): Day to confirm biochemical pregnancy.

On day 15 after embryo transfer, subjects will have a routine pregnancy test (serum  $\beta$ -hCG) to confirm subject's pregnancy. If the test is positive, luteal support is continued up to week 10 of the pregnancy (week 12 gestation).

If pregnancy is not confirmed on Visit 4 the early discontinuation visit should be performed including physical examination and vital signs. Blood samples will be taken for routine laboratory values.

Visit 5 (Day 43 +/- 3 days – Week 6): Day to confirm ongoing pregnancy

Study medication packages should be returned. If pregnancy is confirmed according to clinical evidence then the new study medication packages will be dispensed. Pregnancy related TEAEs and concomitant medication will be recorded.

If an event of miscarriage occurs between the Visits 4 and 6, patient should return to the study site for the early discontinuation visit within 30 days of the last treatment dose or keep their appointment for Visit 6, whatever occurs first. A physical examination including vital signs will be performed; blood samples will be taken for routine laboratory values. Concomitant medication and any TEAEs will be recorded; the patient will return the remaining study medication.

- Visit 6 (Day 71 +/- 3 days Week 10 [12 weeks of gestation]): End of treatment A transvaginal ultrasound examination will be performed to establish an ongoing pregnancy defined as the presence of fetal heart beats. Data on vital signs, routine laboratory values, TEAEs, and concomitant medication will be recorded. Patients return their study medication.
- Visit 7 and 8 (Day 101 +/- 3 days and Day 157 +/- 3 days): Post treatment surveillance calls

Subjects will be followed during the pregnancy by routine pregnancy supervision program until the date of delivery. In addition 2 telephone calls (on Day 101 +/- 3 days and on Day 157 +/- 3 days) will be done to record any concomitant treatment and medications and any TEAEs. Especially events of miscarriage and preterm delivery will be recorded.

- Visit 9: After successful delivery

The time of delivery (gestational age) and the following parameters of the newborn(s) will be obtained: gender, APGAR Score, weight, height, head circumference, abnormal findings of physical examination.

- Visit 10 (Day 30 +/- 3 days after delivery or end of treatment): A phone call will be performed to record both mother' and newborn's safety and wellbeing.

#### 3.2 Study Flowchart

The flowchart of the study can be found in Appendix 9.1.

#### 3.3 Study Objectives

#### **Primary Efficacy Objective(s):**

The primary objective is to demonstrate non-inferiority of the oral dydrogesterone treatment versus the comparator micronized progesterone vaginal gel. The primary efficacy parameter is the pregnancy rate defined as the presence of fetal heart beats at 12 weeks gestation (10 weeks pregnancy) determined by transvaginal ultrasound.

#### **Secondary Efficacy Objective(s):**

The secondary objectives and parameters are a positive pregnancy test on Day 15 after embryo transfer and the incidence of live births and healthy newborns.

#### **Safety Objective(s):**

The safety objective is to obtain safety and tolerability data by means of documentation of treatment emergent adverse events (TEAEs) during the entire study period. In addition, data on vital signs, physical examination findings, and routine laboratory values will be obtained. Furthermore, signs and symptoms of threatened abortion will be recorded. The time of delivery (gestational age) and the following parameters of the newborn will be obtained at delivery: gender, APGAR Score, weight, height, head circumference, abnormal findings of physical examination and any malformations.

#### 3.4 Sample Size and Randomization

Assuming a 35% pregnancy rate for the dydrogesterone and the micronized progesterone gel group, a sample size of about 479 patients per group will provide 90% power to reject the null hypothesis of  $H_0$ :  $p_{dupha} - p_{crinone} \le -0.1$  in favor of the alternative:  $H_1$ :  $p_{dupha} - p_{crinone} \ge -0.1$  with a one sided significance level of 2.5%.

Assuming a dropout rate of 10%, a total sample size of 533 subjects per treatment group will be required, resulting in a total sample size of 1066 subjects in order to show non inferiority in the primary efficacy parameter.

Subjects will be assigned to a treatment group using a centralized electronic system (interactive web response system; IWRS/IRT). The IWRS/IRT assigns a 5-digit randomization number to each subject. Subjects will be allocated in a 1:1 ratio of both treatments in blocks of 4 subject numbers per block. Randomization will be stratified by age group (< 35 years, >= 35 years) and country.

#### 4. STATISTICAL ANALYSIS

## 4.1 Subject samples

There will be six subject samples.

The Re-Randomized subject sample will consist of all subjects who:

- gave their informed consent
- have been randomized for this study before and are re-randomized
- have been allocated to treatment

The All Subjects Consented subject sample will consist of all subjects who:

- gave their informed consent.
- are not included in the Re-Randomized subject sample. All screen failures are kept regardless if they were re-screened or re-randomized.

The All Subjects Allocated to Treatment subject sample will consist of all subjects who:

- are in the All Subjects Consented sample
- were allocated to treatment.

The Safety subject sample will consist of all subjects who:

- are in the All Subjects Allocated to Treatment subject sample
- received at least one dose of study medication.

The Full Analysis (FA) subject sample will consist of all subjects who:

- are included in the Safety subject sample
- had a successful embryo transfer performed at Visit 3 (Day 3 to 6) or prematurely discontinued prior to embryo transfer at Visit 3 (Day 3 to 6) due to study drug related issues, which means that an AE with causality "possible" or "probable" leading to study termination was reported. (Those subjects that discontinued prematurely due to reasons independent of study drug do not contribute to the treatment effect assessment because they did not get an embryo transfer and, therefore, could not get pregnant in their cycle, and the reason for that had nothing to do with any sort of treatment effect).

The Per Protocol (PP) subject sample will be defined through blind data review and will consist of all subjects who:

- are included in the Full Analysis sample
- did not present any major protocol deviations
- had a successful embryo transfer at Visit 3 (Day 3 to 6)

## 4.2 Efficacy analysis

The FA and the PP subject samples will be used for the analysis of the efficacy data. The primary efficacy analysis is to be performed on the PP subject sample (in line with the objective of non-inferiority) and repeated for the FA subject sample. Further statistical tests will be performed, also on secondary variables. All efficacy parameters will be summarized by standard descriptive methods.

The following subgroups are defined for key efficacy analyses:

Age Group:

- < 35 Years
- $\rightarrow = 35 \text{ Years}$

Age (Years) is calculated relative to Screening.

Country:

- Australia
- Belgium
- China
- Germany
- Hong Kong
- India
- Russia
- Singapore
- Thailand
- Ukraine

Baseline BMI (kg/m2):

- < 24
- >= 24 to < 28
- >= 28

Number of embryos transferred:

- One
- Two
- Three

Race:

- Asian
- White

- Other (American Indian or Alaskan Native, Black, of African heritage or African American, Native Hawaiian or Other Pacific Islander)

Weight at baseline:

- < 55 kg
- 55 < 65 kg
- 65 < 75 kg
- >= 75 kg

#### **4.2.1** Calculation of Pregnancy Rates

Denominator

FA subject sample: The rates for the efficacy variables are calculated relative to the number of subjects who:

- Received at least one administration of study drug.
- Had a successful embryo transfer performed at Visit 3 (Day 3 to 6) or prematurely discontinued prior to embryo transfer at Visit 3 (Day 3 to 6) due to study drug related issues.

PP subject sample: The rates for the efficacy variables are calculated relative to the number of subjects who:

- Received at least one administration of study drug.
- Had a successful embryo transfer performed at Visit 3 (Day 3 to 6).
- Did not present any major protocol deviations
- Numerator

A detailed list of subjects who prematurely discontinued, with reasons for discontinuation will be used in the BDR meeting in order to decide which subjects can be included as successes or failures (i.e. not pregnant at Visit 6 (Week 10)).

The numerator for the pregnancy rates will consist of the following subjects counted as successes or failures:

| | After a pregnancy test was performed | |
|---|---|---|
| Pregnancy | Subjects counted as success if: | Subjects counted as failures if: |
| Test | | |
| β-HCG<br>(Visit 4) | Pregnant at Visit 4 (Day 17 to 20) (if the serum \( \beta\)-HCG test is positive the subject will be counted as pregnant) Only for PP: No additional Progesterone was given before visit 4. | Not pregnant at Visit 4 (Day 17 to 20) or ß-HCG test assessments or results is missing (due to test being not performed or subject discontinued prior to visit 4) Only for PP: Additional Progesterone was given before visit 4. |
| Ultrasound<br>(Visit 6) | Pregnant at Visit 6 (Week 10) (gestational sac with viable fetal heart beats) Only for PP: No additional Progesterone was given before visit 6. Pregnancy Status at Visit 5 (Week 6) carr - Data for Visit 6 (Week 10) not avail | Not pregnant at Visit 6 (Week 10) Only for PP: Additional Progesterone was given before visit 6. |
| | Pregnant at Visit 5 (Week 6) and no discontinuation data as in right column present Pregnancy Status at Visit 4 (Day 17 to 20) Data for Visit 5 (Week 6) and Visit | <ul> <li>Not pregnant at Visit 5 (Week 6)</li> <li>Subject prematurely discontinued after Visit 4 (Day 17 to 20) or Visit 5 (Week 6) due to an AE Subject prematurely discontinued after Visit 4 (Day 17 to 20) or Visit 5 (Week 6) with reason of lack of efficacy</li> <li>Only for PP: <ul> <li>Additional Progesterone was given before visit 5</li> </ul> </li> <li>ocarried forward if:</li> </ul> |
| | Pregnant at Visit 4 (Day 17 to 20) and no discontinuation data as in right column present | <ul> <li>Not pregnant at Visit 4 (Day 17 to 20)</li> <li>Subject prematurely discontinued after Visit 4 (Day 17 to 20) due</li> </ul> |



- Subject prematurely discontinued after Visit 4 (Day 17 to 20) with reason of lack of efficacy or pregnancy not confirmed at Visit 4 (Day 17 to 20)

Only for PP:

Additional Progesterone was given before visit 4.

- Subject who prematurely discontinued after Visit 4 (Day 17 to 20) or Visit 5 (Week 6) with reasons, "withdrawal of consent, administrative, lost to follow up and protocol violation" will be discussed on a case by case basis during the BDR meeting.
- For each subject, the reason for premature discontinuation, the time point and any further information will be discussed during the BDR meeting to decide whether the subjects can be counted as a failure or success in the primary analysis.
- The results of the final BDR indicated no such cases to decide on.

## 4.2.2 Primary Efficacy Analysis

The primary efficacy parameter is the comparison of ongoing pregnancy rates, defined as the presence of fetal heart beats at 12 weeks gestation by transvaginal ultrasound. The primary efficacy analysis is using a two-sided 95% confidence interval with a non-inferiority margin of 10% for the difference in pregnancy rates in the two treatment groups.

A non-inferiority margin of 10% was chosen based on data from the previously approved Lutinus®/Endometrin® drug.

The following hypotheses are tested at a one-sided significance level of 2,5%:

- $H_0$ :  $p_{dupha} p_{crinone} \le -\Delta$
- $H_1$ :  $p_{dupha} p_{crinone} > -\Delta$

with  $p_{dupha}$  and  $p_{crinone}$  as the probabilities of pregnancy under Duphaston treatment and Crinone, respectively, and  $\Delta$ =10% as the clinically non-relevant difference accepted as the lower bound of non-inferiority. In order to calculate the confidence intervals, a Cochran-Mantel-Haenszel test stratified for country and age groups will be used (randomization was stratified by country and age group). If Mantel Haenszel estimators cannot be computed, since not both treatment groups are present for an age group in a specific country, the test will only be stratified by age group. The two age groups were defined as patients either older or younger than 35 years. Mantel-Haenszel estimators  $\vec{d}_{MH}$  for the differences of proportions using Cochran's weights are defined as:

$$\widehat{d}_{MH} = \left(\sum_{h} \widehat{d}_{h} w_{h}\right) / \left(\sum_{h} w_{h}\right)$$

with  $\hat{d}_h = \hat{p}_{dupha,h} - \hat{p}_{crimone,h}$  the risk difference in stratum h,  $w_h = n_{dupha,h} * n_{crimone,h}/n_h$  the weight in stratum h and  $n_h$  the number of patients in stratum h. The variance of each stratum specific proportion difference  $p_{dupha} - p_{crinone}$  will be estimated as

$$\hat{p}_{dupha}(1 - \hat{p}_{dupha})/n_{dupha} + \hat{p}_{crinone}(1 - \hat{p}_{crinone})/n_{crinone}$$
.

Assuming that  $\vec{d}_{MH}$  is normally distributed by approximation,  $(\vec{d}_{MH} \pm (z_{1-\alpha/2} * \sigma(\vec{d}_{MH})/\sqrt{n}))$  is the 95% confidence interval for the difference of pregnancy rates in each treatment group (with alpha=5%), which will be compared to  $\Delta$ . In order to declare non-inferiority, the lower bound of the two-sided 95% confidence interval, actually the 97.5% lower confidence bound, should exclude a difference greater than 10% in favor of Duphaston. When that is the case H<sub>0</sub> can be rejected. Since no multiple testing is performed, the type I error alpha does not have to be adjusted.

If the null hypothesis of inferiority can be rejected, a second hypothesis of superiority will be tested with the following hypothesis:

- $H_0$ :  $p_{dupha} p_{crinone} \le 0$
- $H_1$ :  $p_{dupha} p_{crinone} > 0$

To show superiority the lower bound of the 95% confidence interval calculated above should be greater than 0%, for  $H_0$  to be rejected. If non-inferiority can not be established, no further test for superiority will be conducted.

The p-value will be computed for the non-inferiority and if applicable for the superiority test.

The p-value for the hypothesis of non-inferiority is defined as  $P(\hat{d}_{MH} \ge d)$ , with d being the realization of  $\hat{d}_{MH}$  given the specific data, under the assumption that  $H_0$  is correct. Since the normal distribution is invariant under linear transformations,

 $\hat{d}_{MH}/\hat{\sigma}(\hat{d}_{MH})$  is standard normally distributed. Therefore the p-value can be written as

$$1 - \phi \left( \frac{\hat{d}_{\mathit{MH}} + \Delta}{\hat{\sigma}(\hat{d}_{\mathit{MH}}) / \sqrt{n}} \right)$$

Point estimate and 95% confidence intervals for each treatment group separately will be displayed for each rate separately. These confidence intervals are not stratified.

Subgroup analyses:

The primary analysis will be repeated for each of the subgroups defined.

## 4.2.3 Secondary efficacy analysis

The secondary efficacy parameters analyzed are:

- chemical pregnancy rate ( $\beta$ -HCG test) on Day 15 after embryo transfer
- pregnancy rate at visit 5
- biochemical pregnancy rate
- abortion and preterm birth rates
- incidence of live birth and healthy newborns
- gestational age

Gestational age is derived as (date of birth - date of embryo transfer +1day) /7 + 2 weeks. It will be presented in weeks, rounded to two decimal points.

For the calculation of abortion, preterm birth and biochemical rates derived variables will be used instead of qualitative CRF data .A pregnancy outcome is defined as an abortion if the pregnancy is ongoing at visit 5 and gestational age is <= 22 weeks.

Preterm birth is defined as a pregnancy outcome with gestational age greater 22 weeks and less than 37 weeks. Pregnancy outcomes with gestational age >= 37 weeks will be counted as birth. The pregnancy outcome is defined as biochemical pregnancy for all subjects who have an AE "biochemical pregnancy".

The rates for the efficacy variables are calculated relative to the number of subjects who had an embryo transfer done at Visit 3 (Day 3 to 6).

The following parameters of the newborn will be analyzed:

- APGAR score, as well as gender, height, weight and head circumference.
- any malformations and abnormal findings of a physical examination of the newborn.

For the pregnancy rate as well as the rates of live births and healthy newborns p-values will be computed using the same method as for the primary analysis. For the abortion, preterm birth and biochemical pregnancy rates p-values will be calculated with the same methods for the following hypothesis of non-inferiority:

- $H_0$ :  $p_{crinone} p_{dupha} \le -\Delta$
- $H_1$ :  $p_{crinone} p_{dupha} > -\Delta$

The point estimate and 95 % confidence interval (using the stratified CMH approach) for the difference in treatment group for each of the following variables will be presented graphically using forest plots:

- Pregnancy rate (Ultrasound) at visit 6
- Pregnancy rate (β-HCG) at visit 4
- Pregnancy rate at visit 5
- Biochemical pregnancy rate
- Abortion rate
- Preterm birth rate

- Live birth rate (sum of pre-term births and births)
- Healthy newborn rate

Subjects who give birth to more than one healthy newborn will be counted only once.

For each treatment group all efficacy parameters will be summarized by standard descriptive methods.

#### 4.2.4 Other efficacy analysis

For the Chinese sub-report the efficacy analysis will be performed on specifically defined patients. Outputs will be produced for all patients from Chinese sites, Asian sites (which include China, Hong-Kong, India, Singapore and Thailand) and for all patients of Asian race respectively. The analysis is the same as described for the primary and secondary variables.

## 4.3 Safety analysis

The Safety subject sample will be used for the analysis of the safety and tolerability data. The safety and tolerability data collected during this study includes vital signs, routine laboratory values and adverse events. Safety variables will be summarized by standard descriptive statistics.

The baseline period will be defined as the period from informed consent to the first study drug administration. The baseline value for a variable is defined as the last non-missing value collected before first study drug administration. This first day of drug administration is referred to as Day 1. All assessment dates will be related to the first day of study drug administration.

A gap period of infinity will be defined for all safety variables.

#### Adverse Events:

An AE that starts during a unique treatment or that already exists before the start of that unique treatment but worsens during the treatment, including any subsequent wash-out or post-treatment period will be considered as treatment emergent for that unique treatment.

For the definition of treatment emergent, the following unique treatments are distinguished by applicable study period:

- 30 mg dydrogesterone (Duphaston)
- 8% micronized progesterone gel 90 mg (Crinone)

AEs will be reported on a per-subject basis, i.e. counting subjects rather than events. This means that if a subject suffers the same AEs repeatedly during the applicable study period, the event will be counted only once for that period. Repeated events per subject will be summarized according to the following rule: if a subject suffered the same AE more than once, the event will be assigned the worst severity, the closest relationship to the study drug and the earliest starting date. Only treatment emergent AEs will be reported. In the listings, however, all occurrences of the AEs will be presented.

For each unique treatment, treatment emergent AEs will be summarized per primary SOC, per HLT by primary SOC and per PT by HLT and primary SOC. Severity and drug-event relationship of treatment emergent AEs are summarized separately.

Adverse Events are recorded for the mother and the foetus/newborn and will be analyzed separately.

Adverse Events of special interest include: Preterm Birth, Abortion/Miscarriage, Signs and Symptoms of Threatened Abortion.

Adverse Events of Special Interest by Visit Interval include but are not limited to: Abortion, Miscarriage and Malformations.

Adverse Events are coded using Medical Dictionary for Regulatory Activities (MedDRA) version 18.1.

For the Chinese sub-report some tables and listings will also be produced for all patients from Chinese sites, Asian sites and for all patients of Asian race respectively.

#### Vital Signs:

Vitals signs, including changes from baseline will be summarized for baseline, visit 6 and end of treatment. End of treatment is the last assessment (scheduled or unscheduled) and includes data from patients who had the vital signs assessment at their early discontinuation visit. A frequency table will be presented for markedly abnormal values.

Height and weight must be recorded during the treatment phase.

Systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate are to be measured while the subject is in sitting position after 3-5 minutes rest.

#### **Routine Laboratory:**

Laboratory variables, including changes from baseline will be summarized for baseline, visit 6 and end of treatment. End of treatment is the last assessment (scheduled or unscheduled) and includes data from patients who had the laboratory assessment at their early discontinuation visit. A frequency table will be presented for markedly abnormal values. Shift tables will be presented according to the reference ranges (low, normal or high).

Blood will be collected for the determination of the following parameters: Baseline routine laboratory values (hematology: hemoglobin, hematocrit, RBC count, WBC count, platelet count; biochemistry: glucose (if possible fasting), creatinine, alkaline phosphatase, total bilirubin, ALAT, ASAT, gamma-glutamyl transferase, uric acid, calcium, phosphate and potassium.

Urine analysis: Urine sample collection for routine urine analysis of pH, nitrite, specific gravity, blood, protein and glucose will be performed, as well as for pregnancy test (strip test).

For values outside the normal range (or abnormal results) the clinical significance is to be judged by the Investigator.

#### Physical Examination:

A physical examination should be performed and any relevant findings are to be recorded on the Medical History form in the case report form (CRF) (for findings from the past that occurred prior to first screening visit), or on the Adverse Events form in the CRF for findings presently occurring.

## 4.4 Interim Analysis

No interim analysis is planned.

## 4.5 Data Safety Monitoring Board

Not applicable.

## 4.6 Safety Management Team

Not applicable.

# 5. DESCRIPTION OF NON-STANDARD DATA COLLECTED AND DERIVED VARIABLES

#### 5.1 Other Non-Standard Baseline Characteristics

Not applicable.

#### 5.2 Non-Standard Disease History

For the non-standard disease history the number of previous IVF attempts in the subject's life and for this child wish are recorded.

## 5.3 Efficacy data

The following non-standard efficacy parameters are analyzed:

- pregnancy rate (transvaginal ultrasound)
- chemical pregnancy rate (β-HCG test) on Day 15 after embryo transfer
- abortion rate
- biochemical pregnancy rate
- preterm birth rate
- live birth rate
- healthy newborn rate
- gestational age

The following non-standard efficacy data are collected on the newborn:

- Gender:
  - Male
  - Female
- Height at birth (cm)
- Weight at birth (g)
- Head circumference at birth (cm)
- Abnormal findings of physical examination:
  - Yes/Specifications
  - No
- Malformations:
  - Yes/Specifications
  - No
- APGAR score:
  - 1 min postpartal

#### - 5 min postpartal

Newborn efficacy data recorded on the "Status at End of Pregnancy" form will be summarized using descriptive statistic displaying mean, SD, median, min and max values for each applicable safety variable. For qualitative newborn efficacy data, per category the number and frequencies of newborns with non-missing data (n, %) will be the default summary presentation. This data will also be presented in a listing.

#### 5.4 Non-standard Safety Data

Not applicable.

#### 5.5 Drug Accountability and Exposure

#### 5.5.1 Drug Accountability

Treatment compliance/drug accountability is defined as the number of tablets/gel applicators that were actually taken relative to the number of tablets/gel applicators that should have been taken for the duration of actual treatment exposure.

The overall compliance, assessed by tablet/gel applicator count, will be calculated as follows:

Interval Treatment Duration = (Dispensing Date at end of interval – (Dispensing Date at start of interval + 1 day))+1. For the first interval first day of study drug is used as start of interval and for the last interval last day of study drug is used as end of interval.

Overall Treatment Duration = (Last day of study drug administration – First day of study drug administration) + 1.

The calculated percentage compliance will be categorized as:

- Too Low: < 80% compliance.
- Adequate:  $\geq 80\%$  to  $\leq 120\%$  compliance.
- Too High: > 120% compliance.

#### 5.5.2 Exposure

Exposure duration to treatment is equal to the day number of the last day of drug administration, calculated relative to the start of study drug administration.

| Scheduled Treatment Duration Per Treatment Group (Days) | | |
|---|---|---|
| Visit Interval | Duphaston | Crinone |
| Visit 2 to<br>Visit 4 | 17 to 20 | 17 to 20 |
| Visit 4 to<br>Visit 5 | 21 to 30 | 21 to 30 |

| Visit 5 (Week 6) to<br>Visit 6 (Week 10) | 29 | 29 |
|------------------------------------------|----|----|
| Overall | 71 | 71 |

# 6. FURTHER SPECIFICATIONS TO THE STANDARD ANALYSES IN MODULE 2

## 6.1 Trial Design [2]

#### **6.1.1** Trial Periods

The combination of trial arms and trial periods for the current trial is presented in the following diagram:

| Treatment Arm | Screening<br>Period | Treatment<br>Period | Follow-up Period |
|---|---|---|---|
| Duphaston | Amendment1 1-14 days Amendment2 1-40 days | 70 days (+/- 3 days) | From visit 6 (end of treatment period or early discontinuation) until visit 10 (30 days after end of treatment or after delivery) |
| Crinone | Amendment1 1-14 days Amendment2 1-40 days | 70 days (+/- 3 days) | From visit 6 (end of treatment period or early discontinuation) until visit 10 (30 days after end of treatment or after delivery) |

#### Screening Period

Screening period is defined as the period from informed consent to randomization and first study drug administration at Day 1.

#### **Treatment Period**

Treatment period is defined as the period from first dose of study drug at Visit 2 up to and including last day of study drug at Visit 6 or early discontinuation.

#### Follow-up Period

The follow-up period consists of Visits 6 to 10. Visits 7 and 8 are post treatment surveillance calls, which take place every two months. Visit 7 will be at Day 101 (+/- 3 days) and Visit 8 at Day 157 (+/- 3 days). Visit 9 will be performed after delivery, if applicable. Visit 10 is the final follow-up call 30 days after delivery or end of treatment.

#### **6.1.2** Trial Elements

The start time of each intervention will be expressed relative to the first administration of investigational study drug closest to that intervention.

The Trial Elements are presented in the following diagram:

| Trial<br>Element | Description of<br>Element | Rule for Start of<br>Element | Rule for End of<br>Element | Planned<br>Duration of<br>Element |
|---|---|---|---|---|
| SCRN | Screening | Informed consent | Day before first<br>dose of<br>randomized<br>treatment | Amendment1 up to 14 days Amendment2 up to 40 days |
| Duphaston | Dydrogesterone 30 mg daily | Day of first dose of Duphaston | Day of last dose of Duphaston | 70 (+/- 3 days) |
| Crinone | Intravaginal progesterone gel 90 mg daily | Day of first dose of Crinone | Day of last dose of Crinone | 70 (+/- 3 days) |
| FU | Follow-up | End of treatment or early discontinuation | 30 Days after<br>end of treatment<br>or delivery | |

#### 6.1.3 Trial Arms

The trial arms for this study are made up of the following trial elements:

| | Elements | | |
|-----------|----------|-----------|----|
| Trial Arm | | | |
| Duphaston | SCRN | Duphaston | FU |
| Crinone | SCRN | Crinone | FU |

### **6.1.4** Unique Treatments

The trial arms for this study are made up of the following unique treatments:

| Unique treatn | nent | Arm | Elements |
|---------------------|-------|-----------|-----------|
| Description | Label | | |
| Duphaston Duphaston | | Duphaston | Duphaston |
| Crinone Crinone | | Crinone | Crinone |

#### 6.1.5 Visits and related definitions

Tests and examinations that were scheduled in the protocol will be related to the general time axis of the trial by relating the visit date on which a test or examination is performed to the start date of the trial element that describes the first administration of investigational study drug closest in time to the visit date of that test or examination (Reference Start Date/ Time).

| Test /<br>Examination | Visit name | Visit Label | Visit<br>Number | Reference<br>Start<br>Date/Time | Relative Day<br>Number |
|---|---|---|---|---|---|
| See App. 9.1 | Visit 1 | Screening | 1 | | Amendment1 |
| | (Screening and Enrollment) | | | | -14 to -1 |
| | | | | | Amendment 2 |
| | | | | | -40 to -1 |
| See App. 9.1 | Visit 2 (Start of treatment/ Day of oocyte retrieval) | Start of treatment | 2 | Date of first<br>dose of study<br>medication | 1 |
| See App. 9.1 | Visit 3 (Day of embryo transfer (ET)) | Embryo<br>transfer | 3 | Date of first<br>dose of study<br>medication | 3 to 6 |
| See App. 9.1 | Visit 4 (Day to confirm biochemical pregnancy) | Biochemical pregnancy | 4 | Date of first<br>dose of study<br>medication | 17 to 20 |
| See App. 9.1 | Visit 5 (Day to confirm ongoing pregnancy) | Ongoing pregnancy | 5 | Date of first<br>dose of study<br>medication | 43 (+/- 3) |
| See App. 9.1 | Visit 6 (End of treatment/ early discontinuation) | End of treatment | 6 | Date of first<br>dose of study<br>medication | 71 (+/- 3) |
| See App. 9.1 | Visit 7 (Post<br>treatment<br>surveillance<br>call) | First phone call | 7 | Date of first<br>dose of study<br>medication | 101 (+/- 3) |
| See App. 9.1 | Visit 8 (Post<br>treatment<br>surveillance<br>call) | Second phone call | 8 | Date of first<br>dose of study<br>medication | 157 (+/- 3) |
| See App. 9.1 | Visit 9 (After delivery case notes) | After delivery | 9 | | |
| See App. 9.1 | Visit 10 (Phone call 30 days | Final phone call | 10 | Date of | 30 |

| after delivery) |
|-----------------|

## **6.2** Further Specifications to the Standard Tables in Module 2

Not applicable

## 6.3 Other Further Specifications

Not applicable.

#### 7. CHANGES TO PLANNED ANALYSES

## 7.1 Changes to the Analysis as Laid Down in the Protocol

For the subgroup analysis baseline BMI is used instead of baseline weight to align analysis with LOTUS I. Number of embryos transferred was added as a further subgroup. In the protocol of study M13-625 it is mentioned that the day of first study drug administration is Day 0. In this SAP the day of first study drug administration will be defined as Day 1.

Subjects are only included in the study with their first attempt. A sixth subject sample (Re-Randomized subject sample) is introduced consisting of all subjects who gave their informed consent and have been randomized for this study before. The all subject consented subject sample will only consist of patients who gave their informed consent and have not been randomized for this study before. Only demography and AEs listings will be produced for the Re-Randomized subject sample, the data will not be analyzed. Data from re-randomized patients that are screening failures will not be listed or analyzed. Gestational Age will be derived instead of using recorded pregnancy week + 2 weeks.

#### 7.2 Changes from SAP Version 2.0 to Version 3.0

No changes will be made to the final SAP, Version 3.0. If the actual analysis deviates from the final planned analysis, this will be discussed in the Clinical Study Report.

31

#### 8. REFERENCE

- 1. Abbott SAP Module 2
- 2. CDISC terminology, see http://www.cdisc.org.

## 9. APPENDICES

## 9.1 Study Flowchart

| Period | Screening<br>and<br>Enrollment | Start of<br>treatment<br>Day of<br>oocyte<br>Retrieval | Day of<br>embryo<br>transfer<br>(ET) | Day to<br>confirm<br>biochemical<br>pregnancy | Day to<br>confirm<br>ongoing<br>pregnancy | End of<br>Treatment/<br>Early<br>discontinuation* | Post<br>treatment<br>surveillance<br>calls every 2<br>months | After<br>delive<br>ry<br>Case<br>notes | Phone<br>call 30<br>days<br>after<br>delivery |
|---|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4** | 5 | 6 | 7 + 8 | 9 | 10 |
| Day | -40 to -1 | 1 | 3 to 6 | 17 to 20 | 43 (+/- 3 days) | 71 (+/- 3 days) | 101 (+/- 3 days)<br>157 (+/- 3 days) | | |
| Informed consent | X | | | | | | | | |
| Demographic data | X | | | | | | | | |
| Medical history | X | | | | | | | | |
| Physical examination | X | | | | | X | | | |
| Transvaginal ultrasound examination | X | | | | | X should not be performed at the early discontinuation visit | | | |
| Inclusion/exclusion criteria* | X | | | | | | | | |
| Blood samples for routine laboratory values | X | | | | | X | | | |
| β-HCG Test | | | | X | | | | | |
| Urine analysis HCG test (strip test) | X | | | X<br>X | | X | | | |
| Vitals signs | X | | | | | X | | | |

| Period | Screening<br>and<br>Enrollment | Start of<br>treatment<br>Day of<br>oocyte<br>Retrieval | Day of embryo transfer (ET) | Day to confirm biochemical pregnancy | Day to confirm ongoing pregnancy | End of<br>Treatment/<br>Early<br>discontinuation* | Post<br>treatment<br>surveillance<br>calls every 2<br>months | After<br>delive<br>ry<br>Case<br>notes | Phone call 30 days after delivery |
|---|---|---|---|---|---|---|---|---|---|
| Subject to collect<br>study drug at<br>pharmacy | | X | | X | X | | | | |
| Return unused medication | | | | X | X | X | | | |
| Concomitant medication | X | X | X | X | X | X | X | | X |
| Compliance check | | | | X | X | X | | | |
| Adverse events | | X | X | X | X | X | X | X | X |
| Infant assessment***: gender, weight/ height, APGAR, physical examination | | | | | | | | X | |

<sup>\*</sup>For subjects where the hormones values are not available prior screening a hormone testing including FSH, estradiol (E<sub>2</sub>), LH (luteinizing hormone), PRL(Prolactin), T (testosterone) and TSH (thyroid-stimulating hormone) should be performed.

<sup>\*\*</sup>if pregnancy is not confirmed on visit 4 an early discontinuation should be performed including physical examination and blood sampling for routine laboratory testing

<sup>\*\*\*</sup> If an event of miscarriage occurs between the Visits 4 and 6, patient should be return to the study site for the early discontinuation visit within 30 days of the last treatment dose or on their appointment for Visit 6, whatever occurs first. A physical examination including vital signs will be performed; blood samples will be taken for routine laboratory values

<sup>\*\*\*\*</sup> After successful delivery, the time of delivery (pregnancy week) and the following parameters of the newborn baby will be obtained: gender, APGAR score, weight, height, physical examination.

# 9.2 Tables, Listings and Figures

## **9.2.1** Tables

For the shells of the non-standard tables, see Section 10.1.

| | | | | Produced for: |
|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results |
| DST001 | Subject Disposition | 10.1.1.1.1 | Subject Disposition - All Subjects Allocated to Treatment Subject Sample | х |
| DST001 | Subject Disposition | 10.1.1.1.1 | Subject Disposition: Chinese Sites - All<br>Subjects Allocated to Treatment Subject<br>Sample | |
| DST001 | Subject Disposition | 10.1.1.1.2 | Subject Disposition: Asian Sites - All Subjects<br>Allocated to Treatment Subject Sample | |
| DST001 | Subject Disposition | 10.1.1.1.3 | Subject Disposition: Asian Race - All Subjects<br>Allocated to Treatment Subject Sample | |
| DST001 | Subject Disposition | 10.1.1.1.2 | Subject Disposition by Country - All Subjects<br>Allocated to Treatment Subject Sample | |
| DST001 | Subject Disposition | 10.1.1.1.3 | Subject Disposition by Age Group - All<br>Subjects Allocated to Treatment Subject<br>Sample | |
| DVT001 | Protocol Deviations | 10.1.1.2 | Major Protocol Deviations – All Subjects<br>Allocated to Treatment Subject Sample | |
| DVT002 | Protocol Deviations | 10.1.1.3 | Subject Samples - All Subjects Allocated to Treatment Subject Sample | х |
| DMT002 | Demographic Data | 10.1.1.4.1 | Demographics – Full Analysis Subject Sample | x |
| DMT002 | Demographic Data | 10.1.1.4.2 | Demographics by Country – Full Analysis<br>Subject Sample | |
| DMT002 | Demographic Data | 10.1.1.4.3 | Demographics- Safety Subject Sample | |
| DMT002 | Demographic Data | 10.1.1.4.3.1 | Demographics: Chinese Sites – Safety Subject<br>Sample | |
| DMT002 | Demographic Data | 10.1.1.4.3.2 | Demographics: Asian Sites – Safety Subject<br>Sample | |
| DMT002 | Demographic Data | 10.1.1.4.3.3 | Demographics: Asian Race – Safety Subject<br>Sample | |
| VST003 | Vital Signs | 10.1.1.5 | Other Baseline Characteristics – Full Analysis<br>Subject Sample | |
| MHT001 | Medical History | 10.1.1.6 | Medical History – Full Analysis Subject<br>Sample | |
| CMT001 | Concomitant<br>Medications | 10.1.1.7 | Concomitant Medication: Subject – Full<br>Analysis Subject Sample | |
| SCT001 | Subject<br>Characteristics | 10.1.1.8 | Number of IVF Attempts – Full Analysis<br>Subject Sample | |
| DAT001 | Treatment<br>Compliance | 10.1.1.8.1 | Compliance to Study Drug – Safety Subject<br>Sample | |

| | | | | Produced for: |
|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results |
| DAT001 | Treatment<br>Compliance | 10.1.1.8.2 | Compliance to Study Drug – Full Analysis<br>Subject Sample | |
| DAT001 | Treatment<br>Compliance | 10.1.1.8.3 | Compliance to Study Drug – Per Protocol<br>Subject Sample | |
| EXT001 | Exposure | 10.1.1.9.1 | Exposure to Study Drug – Safety Subject<br>Sample | |
| EXT001 | Exposure | 10.1.1.9.1.1 | Exposure to Study Drug: Chinese Sites –<br>Safety Subject Sample | |
| EXT001 | Exposure | 10.1.1.9.1.2 | Exposure to Study Drug: Asian Sites – Safety Subject Sample | |
| EXT001 | Exposure | 10.1.1.9.1.3 | Exposure to Study Drug: Asian Race – Safety Subject Sample | |
| EXT001 | Exposure | 10.1.1.9.2 | Exposure to Study Drug – Full Analysis<br>Subject Sample | |
| EXT001 | Exposure | 10.1.1.9.3 | Exposure to Study Drug – Per Protocol<br>Subject Sample | |
| EFT001 | Efficacy | 10.1.2.1.1 | Pregnancy Confirmation at Visit 4 – Full Analysis Subject Sample | х |
| EFT001 | Efficacy | 10.1.2.1.1.1 | Pregnancy Confirmation at Visit 4: Chinese<br>Sites – Full Analysis Subject Sample | |
| EFT001 | Efficacy | 10.1.2.1.1.2 | Pregnancy Confirmation at Visit 4: Asian<br>Sites – Full Analysis Subject Sample | |
| EFT001 | Efficacy | 10.1.2.1.1.3 | Pregnancy Confirmation at Visit 4: Asian Race – Full Analysis Subject Sample | |
| EFT001 | Efficacy | 10.1.2.1.1a | Pregnancy Confirmation at Visit 4 by<br>Country– Full Analysis Subject Sample | |
| EFT001 | Efficacy | 10.1.2.1.1b | Pregnancy Confirmation at Visit 4 by Age<br>Group - Full Analysis Subject Sample | |
| EFT001 | Efficacy | 10.1.2.1.1c | Pregnancy Confirmation at Visit 4 by Race -<br>Full Analysis Subject Sample | |
| EFT001 | Efficacy | 10.1.2.1.1d | Pregnancy Confirmation at Visit 4 by BMI - Full Analysis Subject Sample | x |
| EFT001 | Efficacy | 10.1.2.1.1e | Pregnancy Confirmation at Visit 4 by Number of embryos transferred - Full Analysis Subject Sample | |
| EFT001 | Efficacy | 10.1.2.1.1f | Pregnancy Confirmation at Visit 4 by Weight - Full Analysis Subject Sample | |
| EFT002 | Efficacy | 10.1.2.1.2 | Pregnancy Status at Visit 5 – Full Analysis<br>Subject Sample | х |
| EFT002 | Efficacy | 10.1.2.1.2a | Pregnancy Status at Visit 5 by Country– Full<br>Analysis Subject Sample | |
| EFT002 | Efficacy | 10.1.2.1.2b | Pregnancy Status at Visit 5 by Age Group–<br>Full Analysis Subject Sample | |
| | | | | Produced for: |
|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results |
| EFT002 | Efficacy | 10.1.2.1.2c | Pregnancy Status at Visit 5 by Race– Full<br>Analysis Subject Sample | |
| EFT002 | Efficacy | 10.1.2.1.2d | Pregnancy Status at Visit 5 by BMI – Full<br>Analysis Subject Sample | |
| EFT002 | Efficacy | 10.1.2.1.2e | Pregnancy Status at Visit 5 by Number of<br>embryos transferred – Full Analysis Subject<br>Sample | |
| EFT002 | Efficacy | 10.1.2.1.2f | Pregnancy Status at Visit 5 by Weight – Full<br>Analysis Subject Sample | |
| EFT003 | Efficacy | 10.1.2.1.3 | Pregnancy Status : Transvaginal Ultrasound at Visit 6 – Full Analysis Subject Sample | x |
| EFT003 | Efficacy | 10.1.2.1.3.1 | Pregnancy Status : Transvaginal Ultrasound at<br>Visit 6: Chinese Sites – Full Analysis Subject<br>Sample | |
| EFT003 | Efficacy | 10.1.2.1.3.2 | Pregnancy Status : Transvaginal Ultrasound at<br>Visit 6: Asian Sites – Full Analysis Subject<br>Sample | |
| EFT003 | Efficacy | 10.1.2.1.3.3 | Pregnancy Status : Transvaginal Ultrasound at<br>Visit 6: Asian Race – Full Analysis Subject<br>Sample | |
| EFT003 | Efficacy | 10.1.2.1.3a | Pregnancy Status : Transvaginal Ultrasound at<br>Visit 6 by Country– Full Analysis Subject<br>Sample | X |
| EFT003 | Efficacy | 10.1.2.1.3a. | Pregnancy Status : Transvaginal Ultrasound at<br>Visit 6 by Country: Chinese Sites – Full<br>Analysis Subject Sample | |
| EFT003 | Efficacy | 10.1.2.1.3a.<br>2 | Pregnancy Status : Transvaginal Ultrasound at<br>Visit 6 by Country: Asian Sites – Full<br>Analysis Subject Sample | |
| EFT003 | Efficacy | 10.1.2.1.3a. | Pregnancy Status : Transvaginal Ultrasound at<br>Visit 6 by Country: Asian Race – Full<br>Analysis Subject Sample | |
| EFT003 | Efficacy | 10.1.2.1.3b | Pregnancy Status : Transvaginal Ultrasound at<br>Visit 6 by Age Group– Full Analysis Subject<br>Sample | |
| EFT003 | Efficacy | 10.1.2.1.3c | Pregnancy Status : Transvaginal Ultrasound at<br>Visit 6 by Race– Full Analysis Subject Sample | |
| EFT003 | Efficacy | 10.1.2.1.3d | Pregnancy Status : Transvaginal Ultrasound at<br>Visit 6 by BMI – Full Analysis Subject<br>Sample | |
| EFT003 | Efficacy | 10.1.2.1.3e | Pregnancy Status : Transvaginal Ultrasound at<br>Visit 6 by Number of embryos transferred –<br>Full Analysis Subject Sample | |

| | | | | Produced for: |
|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results |
| EFT003 | Efficacy | 10.1.2.1.3f | Pregnancy Status : Transvaginal Ultrasound at<br>Visit 6 by Weight – Full Analysis Subject<br>Sample | |
| EFT004 | Efficacy | 10.1.2.1.4 | Efficacy Analysis – Full Analysis Subject<br>Sample | X |
| EFT004 | Efficacy | 10.1.2.1.4.1 | Efficacy Analysis: Chinese Sites – Full<br>Analysis Subject Sample | X |
| EFT004 | Efficacy | 10.1.2.1.4.2 | Efficacy Analysis: Asian Sites – Full Analysis<br>Subject Sample | Х |
| EFT004 | Efficacy | 10.1.2.1.4.3 | Efficacy Analysis: Asian Race – Full Analysis<br>Subject Sample | х |
| EFT004 | Efficacy | 10.1.2.1.5 | Efficacy Analysis – Per Protocol Subject<br>Sample | х |
| EFT004 | Efficacy | 10.1.2.1.5.1 | Efficacy Analysis: Chinese Sites – Per<br>Protocol Subject Sample | х |
| EFT004 | Efficacy | 10.1.2.1.5.2 | Efficacy Analysis: Asian Sites – Per Protocol<br>Subject Sample | х |
| EFT004 | Efficacy | 10.1.2.1.5.3 | Efficacy Analysis: Asian Race – Per Protocol<br>Subject Sample | Х |
| EFT004 | Efficacy | 10.1.2.1.4a | Efficacy Analysis by Country– Full Analysis<br>Subject Sample | |
| EFT004 | Efficacy | 10.1.2.1.4b | Efficacy Analysis by Age Group - Full<br>Analysis Subject Sample | |
| EFT004 | Efficacy | 10.1.2.1.4c | Efficacy Analysis by Race – Full Analysis<br>Subject Sample | |
| EFT004 | Efficacy | 10.1.2.1.4d | Efficacy Analysis by BMI – Full Analysis<br>Subject Sample | |
| EFT004 | Efficacy | 10.1.2.1.4e | Efficacy Analysis by Number of embryos transferred – Full Analysis Subject Sample | |
| EFT004 | Efficacy | 10.1.2.1.4f | Efficacy Analysis by Weight – Full Analysis<br>Subject Sample | |
| EFT005 | Efficacy | 10.1.2.1.6 | Gestational Age – Full Analysis Subject<br>Sample | |
| EFT005 | Efficacy | 10.1.2.1.6.1 | Gestational Age: Chinese Sites – Full Analysis<br>Subject Sample | |
| EFT005 | Efficacy | 10.1.2.1.6.2 | Gestational Age: Asian Sites – Full Analysis<br>Subject Sample | |
| EFT005 | Efficacy | 10.1.2.1.6.3 | Gestational Age: Asian Race – Full Analysis<br>Subject Sample | |
| EFT006 | Efficacy | 10.1.2.1.7 | Status at End of Pregnancy: Newborn - Full<br>Analysis Subject Sample | х |
| EFT006 | Efficacy | 10.1.2.1.7.1 | Status at End of Pregnancy: Newborn Chinese<br>Sites - Full Analysis Subject Sample | |

| | | | | Produced for: |
|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results |
| EFT006 | Efficacy | 10.1.2.1.7.2 | Status at End of Pregnancy: Newborn Asian<br>Sites - Full Analysis Subject Sample | |
| EFT006 | Efficacy | 10.1.2.1.7.3 | Status at End of Pregnancy: Newborn Asian<br>Race - Full Analysis Subject Sample | |
| EFT007 | Efficacy | 10.1.2.1.8 | Number of Live Births - Full Analysis Subject<br>Sample | |
| EFT007 | Efficacy | 10.1.2.1.8.1 | Number of Live Births: Chinese Sites - Full<br>Analysis Subject Sample | |
| EFT007 | Efficacy | 10.1.2.1.8.2 | Number of Live Births: Asian Sites - Full<br>Analysis Subject Sample | |
| EFT007 | Efficacy | 10.1.2.1.8.3 | Number of Live Births: Asian Race - Full<br>Analysis Subject Sample | |
| AET001 | Adverse Events | 10.1.3.1.1 | Overall Summary of Adverse Events: Subject - Safety Subject Sample | х |
| AET001 | Adverse Events | 10.1.3.1.1.1 | Overall Summary of Adverse Events: Subject<br>Chinese Sites – Safety Subject Sample | |
| AET001 | Adverse Events | 10.1.3.1.1.2 | Overall Summary of Adverse Events: Subject<br>Asian Sites – Safety Subject Sample | |
| AET001 | Adverse Events | 10.1.3.1.1.3 | Overall Summary of Adverse Events: Subject:<br>Asian Race – Safety Subject Sample | |
| AET001 | Adverse Events | 10.1.3.1.1a | Overall Summary of Adverse Events: Subject by Country– Safety Subject Sample | |
| AET001 | Adverse Events | 10.1.3.1.1b | Overall Summary of Adverse Events: Subject<br>by Age Group– Safety Subject Sample | |
| AET001 | Adverse Events | 10.1.3.1.1c | Overall Summary of Adverse Events: Subject by Race–Safety Subject Sample | |
| AET001 | Adverse Events | 10.1.3.1.1d | Overall Summary of Adverse Events: Subject by BMI– Safety Subject Sample | |
| AET001 | Adverse Events | 10.1.3.1.1e | Overall Summary of Adverse Events: Subject<br>by Number of embryos transferred – Safety<br>Subject Sample | |
| AET001 | Adverse Events | 10.1.3.1.1f | Overall Summary of Adverse Events: Subject by Weight– Safety Subject Sample | |
| AET001 | Adverse Events | 10.1.3.1.2 | Overall Summary of Adverse Events:<br>Newborn – Full Analysis Subject Sample | |
| AET002 | Adverse Events | 10.1.3.1.3 | Incidence of TEAEs – Safety Subject Sample | х |
| AET002 | Adverse Events | 10.1.3.1.3.1 | Incidence of TEAEs: Chinese Sites – Safety Subject Sample | |
| AET002 | Adverse Events | 10.1.3.1.3.2 | Incidence of TEAEs: Asian Sites – Safety<br>Subject Sample | |
| AET002 | Adverse Events | 10.1.3.1.3.3 | Incidence of TEAEs: Asian Race – Safety<br>Subject Sample | |

| | | | | Produced for: |
|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results |
| AET002 | Adverse Events | 10.1.3.1.3a | Incidence of TEAEs by Country – Safety<br>Subject Sample | |
| AET002 | Adverse Events | 10.1.3.1.3b | Incidence of TEAEs by Age Group – Safety<br>Subject Sample | |
| AET002 | Adverse Events | 10.1.3.1.3c | Incidence of TEAEs by Race – Safety Subject<br>Sample | |
| AET002 | Adverse Events | 10.1.3.1.3d | Incidence of TEAEs by BMI - Safety Subject<br>Sample | |
| AET002 | Adverse Events | 10.1.3.1.3e | Incidence of TEAEs by Number of embryos transferred – Safety Subject Sample | |
| AET002 | Adverse Events | 10.1.3.1.3f | Incidence of TEAEs by weight – Safety<br>Subject Sample | |
| AET002 | Adverse Events | 10.1.3.1.4 | Incidence of TEAEs - Newborn – Full<br>Analysis Subject Sample | |
| AET003 | Adverse Events | 10.1.3.1.5 | Incidence of TEAEs in 5% of the Subjects in<br>Any Treatment Group – Safety Subject<br>Sample | |
| AET003 | Adverse Events | 10.1.3.1.5.1 | Incidence of TEAEs in 5% of the Subjects in<br>Any Treatment Group: Chinese Sites – Safety<br>Subject Sample | |
| AET003 | Adverse Events | 10.1.3.1.5.2 | Incidence of TEAEs in 5% of the Subjects in<br>Any Treatment Group: Asian Sites – Safety<br>Subject Sample | |
| AET003 | Adverse Events | 10.1.3.1.5.3 | Incidence of TEAEs in 5% of the Subjects in<br>Any Treatment Group: Asian Race – Safety<br>Subject Sample | |
| AET004 | Adverse Events | 10.1.3.1.6 | Incidence of TEAEs of Special Interest -<br>Safety Subject Sample | |
| AET004 | Adverse Events | 10.1.3.1.6.1 | Incidence of TEAEs of Special Interest:<br>Chinese Sites - Safety Subject Sample | |
| AET004 | Adverse Events | 10.1.3.1.6.2 | Incidence of TEAEs of Special Interest: Asian Sites - Safety Subject Sample | |
| AET004 | Adverse Events | 10.1.3.1.6.3 | Incidence of TEAEs of Special Interest: Asian Race - Safety Subject Sample | |
| AET004 | Adverse Events | 10.1.3.1.6a | Incidence of TEAEs of Special Interest by<br>Country - Safety Subject Sample | |
| AET004 | Adverse Events | 10.1.3.1.6b | Incidence of TEAEs of Special Interest by<br>Age Group - Safety Subject Sample | |
| AET004 | Adverse Events | 10.1.3.1.6c | Incidence of TEAEs of Special Interest by Race – Safety Subject Sample | |
| AET004 | Adverse Events | 10.1.3.1.6d | Incidence of TEAEs of Special Interest by BMI – Safety Subject sample | |

| | | | | Produced for: |
|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results |
| AET004 | Adverse Events | 10.1.3.1.6e | Incidence of TEAEs of Special Interest by<br>Number of embryos transferred - Safety<br>Subject Sample | |
| AET004 | Adverse Events | 10.1.3.1.6f | Incidence of TEAEs of Special Interest by<br>Weight - Safety Subject Sample | |
| AET005 | Adverse Events | 10.1.3.1.7 | Incidence of TEAEs With a Reasonable Possibility for a Causal Relationship (Investigator's Judgment) – Safety Subject Sample | |
| AET005 | Adverse Events | 10.1.3.1.7.1 | Incidence of TEAEs With a Reasonable Possibility for a Causal Relationship (Investigator's Judgment): Chinese Sites – Safety Subject Sample | |
| AET005 | Adverse Events | 10.1.3.1.7.2 | Incidence of TEAEs With a Reasonable Possibility for a Causal Relationship (Investigator's Judgment): Asian Sites – Safety Subject Sample | |
| AET005 | Adverse Events | 10.1.3.1.7.3 | Incidence of TEAEs With a Reasonable<br>Possibility for a Causal Relationship<br>(Investigator's Judgment): Asian Race –<br>Safety Subject Sample | |
| AET006 | Adverse Events | 10.1.3.1.8 | Incidence of TEAEs by Maximum Severity<br>(Investigator's Judgment) – Safety Subject<br>Sample | |
| AET007 | Adverse Events | 10.1.3.1.9 | Incidence of TESAEs: Subject – Safety<br>Subject Sample | |
| AET007 | Adverse Events | 10.1.3.1.9.1 | Incidence of TESAEs: Chinese Sites – Safety Subject Sample | |
| AET007 | Adverse Events | 10.1.3.1.9.2 | Incidence of TESAEs: Asian Sites – Safety<br>Subject Sample | |
| AET007 | Adverse Events | 10.1.3.1.9.3 | Incidence of TESAEs: Asian Race – Safety<br>Subject Sample | |
| AET007 | Adverse Events | 10.1.3.1.9a | Incidence of TESAEs by Country – Safety<br>Subject Sample | |
| AET007 | Adverse Events | 10.1.3.1.9b | Incidence of TESAEs by Age Group – Safety<br>Subject Sample | |
| AET007 | Adverse Events | 10.1.3.1.9c | Incidence of TESAEs by Race - Safety<br>Subject Sample | |
| AET007 | Adverse Events | 10.1.3.1.9d | Incidence of TESAEs by BMI– Safety Subject<br>Sample | |
| AET007 | Adverse Events | 10.1.3.1.9e | Incidence of TESAEs by Number of embryos transferred – Safety Subject Sample | |
| AET007 | Adverse Events | 10.1.3.1.9f | Incidence of TESAEs by Weight – Safety<br>Subject Sample | |

| | | | | Produced for: |
|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results |
| AET007 | Adverse Events | 10.1.3.1.15 | Incidence of TESAEs: Newborn – Full<br>Analysis Subject Sample | |
| AET008 | Adverse Events | 10.1.3.1.10 | Incidence of TEAEs Leading to Study<br>Termination – Safety Subject Sample | |
| AET008 | Adverse Events | 10.1.3.1.10. | Incidence of TEAEs Leading to Study<br>Termination: Chinese Sites – Safety Subject<br>Sample | |
| AET008 | Adverse Events | 10.1.3.1.10. | Incidence of TEAEs Leading to Study<br>Termination: Asian Sites – Safety Subject<br>Sample | |
| AET008 | Adverse Events | 10.1.3.1.10. | Incidence of TEAEs Leading to Study<br>Termination: Asian Race – Safety Subject<br>Sample | |
| AET009 | Adverse Events | 10.1.3.1.11 | Incidence of Non-Serious TEAEs – Safety<br>Subject Sample | |
| AET010 | Adverse Events | 10.1.3.1.12 | Incidence of Non-Serious TEAEs in >= 5% of the Subjects in Any Treatment Group – Safety Subject Sample | |
| AET011 | Adverse Events | 10.1.3.1.13 | Incidence of TEAEs Leading to Discontinuation of Study Drug – Safety Subject Sample | |
| AET0012 | Adverse Events | 10.1.3.1.14 | Adverse Events of Special Interest by Visit<br>Interval – Safety Subject Sample | |
| LBT001 | Laboratory Tests | 10.1.3.2.1 | Summary of Quantitative Safety Laboratory<br>Variables– Safety Subject Sample | |
| LBT002 | Laboratory Tests | 10.1.3.2.2 | Summary of Qualitative Safety Urinalysis<br>Variables– Safety Subject Sample | |
| LBT003 | Laboratory Tests | 10.1.3.2.3 | Shifts of Quantitative Safety Laboratory<br>Variables From Baseline to Each Post-<br>Baseline Visit Based on Reference Ranges –<br>Safety Subject Sample | |
| LBT004 | Laboratory Tests | 10.1.3.2.4 | Incidence of Markedly Abnormal Safety<br>Laboratory Variables – Safety Subject Sample | |
| LBT005 | Laboratory Tests | 10.1.3.2.5 | Changes From Baseline of Qualitative Safety<br>Laboratory Variables – Safety Subject sample | |
| VST001 | Vital Signs | 10.1.3.3.1 | Summary of Vital Signs – Safety Subject<br>Sample | |
| VST002 | Vital Signs | 10.1.3.3.2 | Incidence of Markedly Abnormal Vital Signs - Safety Subject Sample | |

Note: A missing output code denotes a non-standard output.

## 9.2.2 Listings

For the shells of the non-standard listings, see Section 10.2.

| | | | | Produced for: |
|---|---|---|---|---|
| Output | | Output | | Headline |
| Code | Clinical Domain | Number | Title | Results |
| DSL001 | Subject Disposition | 12.2.1.1 | Subjects Who Prematurely Terminated the<br>Study Prior to Treatment Allocation - All<br>Subjects Consented Subject Sample | |
| DSL001 | Subject Disposition | 12.2.1.1.1 | Subjects Who Prematurely Terminated the Study Prior to Treatment Allocation: Chinese Sites - All Subjects Consented Subject Sample | |
| DSL001 | Subject Disposition | 12.2.1.1.2 | Subjects Who Prematurely Terminated the<br>Study Prior to Treatment Allocation: Asian<br>Sites - All Subjects Consented Subject Sample | |
| DSL001 | Subject Disposition | 12.2.1.1.3 | Subjects Who Prematurely Terminated the<br>Study Prior to Treatment Allocation: Asian<br>Race - All Subjects Consented Subject Sample | |
| DSL002 | Subject Disposition | 12.2.1.2 | Subjects Allocated to Treatment - All Subjects<br>Allocated to Treatment Subject Sample | |
| DSL003 | Subject Disposition | 12.2.1.3 | Subjects Allocated to Treatment Who<br>Prematurely Terminated the Study - All<br>Subjects Allocated to Treatment Subject<br>Sample | |
| DSL004 | Subject Disposition | 12.2.1.4 | Subjects Allocated to Treatment Who<br>Prematurely Terminated the Study due to a<br>Protocol Violation- All Subjects Allocated to<br>Treatment Subject Sample | |
| DVL001 | Major Protocol<br>Deviations | 12.2.2.1 | Subjects With Major Protocol Deviations -<br>All Subjects Allocated to Treatment Subject<br>Sample | |
| IEL002 | Inclusion/Exclusion | 12.2.2.2 | Subjects With Deviations from Inclusion or<br>Exclusion Criteria - All Subjects Allocated to<br>Treatment Subject Sample | |
| DVL002 | Major Protocol<br>Deviations | 12.2.2.3 | Subjects Excluded From the Subject Samples -<br>All Subjects Allocated to Treatment Subject<br>Sample | |
| DML002 | Demographic Data | 12.2.4.1 | Demographics - All Subjects Allocated to<br>Treatment Subject Sample | |
| DML002 | Demographic Data | 12.2.4.1.1 | Demographics: Chinese Sites - All Subjects<br>Allocated to Treatment Subject Sample | |
| DML002 | Demographic Data | 12.2.4.1.2 | Demographics: Asian Sites - All Subjects<br>Allocated to Treatment Subject Sample | |
| DML002 | Demographic Data | 12.2.4.1.3 | Demographics: Asian Race - All Subjects<br>Allocated to Treatment Subject Sample | |
| DML002 | Demographic Data | 12.2.4.1a | Demographics – Re-Randomized Subject<br>Sample | |
| VSL003* | Vital Signs | 12.2.4.2 | Other Baseline Characteristics - All Subjects<br>Allocated to Treatment Subject Sample | |

| | | | | Produced for: |
|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results |
| MHL001 | Medical History | 12.2.4.3 | Medical History: General - All Subjects<br>Allocated to Treatment Subject Sample | |
| MHL002 | Medical History | 12.2.4.4 | Medical History: MedDRA Coding - All<br>Subjects Allocated to Treatment Subject<br>Sample | |
| SCL001 | Subject<br>Characteristics | 12.2.4.5 | IVF Attempts – All Subjects Allocated to<br>Treatment Subject Sample | |
| CML001 | Concomitant<br>Medications | 12.2.4.6 | Concomitant Medication: General - All<br>Subjects Allocated to Treatment Subject<br>Sample | |
| CML002 | Concomitant<br>Medications | 12.2.4.7 | Concomitant Medication: Subject: WHO-DD<br>Coding - All Subjects Allocated to Treatment<br>Subject Sample | |
| CML003 | Concomitant<br>Medications | 12.2.4.8 | Concomitant Medication: Newborn – Full<br>Analysis Subject Sample | |
| CML002 | Concomitant<br>Medications | 12.2.4.9 | Concomitant Medication: Newborn: WHO-DD Coding – Full Analysis Subject Sample | |
| DAL001 | Drug Accountability | 12.2.5.1 | Drug Accountability and Compliance - Safety<br>Subject Sample | |
| EFL001 | Efficacy | 12.2.6.1 | Embryo Transfer – Safety Subject Sample | |
| EFL001 | Efficacy | 12.2.6.1.1 | Embryo Transfer: Chinese Sites – Safety<br>Subject Sample | |
| EFL001 | Efficacy | 12.2.6.1.2 | Embryo Transfer: Asian Sites – Safety Subject<br>Sample | |
| EFL001 | Efficacy | 12.2.6.1.3 | Embryo Transfer: Asian Race – Safety Subject<br>Sample | |
| EFL002 | Efficacy | 12.2.6.2 | Pregnancy Confirmation– Full Analysis<br>Subject Sample | |
| EFL002 | Efficacy | 12.2.6.2.1 | Pregnancy Confirmation: Chinese Sites– Full<br>Analysis Subject Sample | |
| EFL002 | Efficacy | 12.2.6.2.2 | Pregnancy Confirmation: Asian Sites– Full<br>Analysis Subject Sample | |
| EFL002 | Efficacy | 12.2.6.2.3 | Pregnancy Confirmation: Asian Race– Full<br>Analysis Subject Sample | |
| EFL003 | Efficacy | 12.2.6.3 | Pregnancy Confirmation: Transvaginal<br>Ultrasound – Full Analysis Subject Sample | |
| EFL003 | Efficacy | 12.2.6.3.1 | Pregnancy Confirmation: Transvaginal<br>Ultrasound: Chinese Sites – Full Analysis<br>Subject Sample | |
| EFL003 | Efficacy | 12.2.6.3.2 | Pregnancy Confirmation: Transvaginal<br>Ultrasound: Asian Sites – Full Analysis<br>Subject Sample | |

| | | | | Produced for: |
|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results |
| EFL003 | Efficacy | 12.2.6.3.3 | Pregnancy Confirmation: Transvaginal<br>Ultrasound: Asian Race – Full Analysis<br>Subject Sample | |
| EFL004 | Efficacy | 12.2.6.4 | Pregnancy Status – Full Analysis Subject<br>Sample | |
| EFL004 | Efficacy | 12.2.6.4.1 | Pregnancy Status: Chinese Sites – Full<br>Analysis Subject Sample | |
| EFL004 | Efficacy | 12.2.6.4.2 | Pregnancy Status: Asian Sites – Full Analysis<br>Subject Sample | |
| EFL004 | Efficacy | 12.2.6.4.3 | Pregnancy Status: Asian Race – Full Analysis<br>Subject Sample | |
| EFL005 | Efficacy | 12.2.6.5 | Status at End of Pregnancy: Subject – Full<br>Analysis Subject Sample | |
| EFL005 | Efficacy | 12.2.6.5.1 | Status at End of Pregnancy: Subject Chinese<br>Sites – Full Analysis Subject Sample | |
| EFL005 | Efficacy | 12.2.6.5.2 | Status at End of Pregnancy: Subject Asian<br>Sites – Full Analysis Subject Sample | |
| EFL005 | Efficacy | 12.2.6.5.3 | Status at End of Pregnancy: Subject Asian<br>Race – Full Analysis Subject Sample | |
| EFL006 | Efficacy | 12.2.6.6 | Status at End of Pregnancy: Newborn – Full<br>Analysis Subject Sample | |
| EFL006 | Efficacy | 12.2.6.6.1 | Status at End of Pregnancy: Newborn Chinese<br>Sites – Full Analysis Subject Sample | |
| EFL006 | Efficacy | 12.2.6.6.2 | Status at End of Pregnancy: Newborn Asian<br>Sites – Full Analysis Subject Sample | |
| EFL006 | Efficacy | 12.2.6.6.3 | Status at End of Pregnancy: Newborn Asian<br>Race – Full Analysis Subject Sample | |
| EFL006 | Efficacy | 12.2.6.7 | Status at End of Pregnancy: Newborn – for<br>Patients from Russia – Full Analysis Subject<br>Sample | |
| EFL009 | Efficacy | 12.2.6.8 | Phone Contacts– Full Analysis Subject<br>Sample | |
| EFL010 | Efficacy | 12.2.6.9 | Final Phone Contact - Full Analysis Subject<br>Sample | |
| AEL008 | Adverse Events | 12.2.7.1 | AEs: General: Subject - All Subjects<br>Consented Subject Sample | |
| AEL008 | Adverse Events | 12.2.7.1a | AEs: General: Subject – Re-Randomized<br>Subject Sample | |
| AEL003 | Adverse Events | 12.2.7.2 | AEs: General: Newborn – Full Analysis<br>Subject Sample | |
| AEL002 | Adverse Events | 12.2.7.3 | AEs: MedDRA Coding - All Subjects<br>Consented Subject Sample | |

| | | | | Produced for: |
|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results |
| AEL002 | Adverse Events | 12.2.7.3.1 | AEs: MedDRA Coding: Chinese Sites - All<br>Subjects Consented Subject Sample | |
| AEL002 | Adverse Events | 12.2.7.3.2 | AEs: MedDRA Coding: Asian Sites - All<br>Subjects Consented Subject Sample | |
| AEL002 | Adverse Events | 12.2.7.3.3 | AEs: MedDRA Coding: Asian Race - All<br>Subjects Consented Subject Sample | |
| AEL002 | Adverse Events | 12.2.7.3a | AEs: MedDRA Coding: - Re-Randomized Subject Sample | |
| AEL002 | Adverse Events | 12.2.7.4 | AEs: MedDRA Coding: Newborn – Full<br>Analysis Subject Sample | |
| AEL002 | Adverse Events | 12.2.7.4.1 | AEs: MedDRA Coding: Newborn Chinese<br>Sites – Full Analysis Subject Sample | |
| AEL002 | Adverse Events | 12.2.7.4.2 | AEs: MedDRA Coding: Newborn Asian Sites - Full Analysis Subject Sample | |
| AEL002 | Adverse Events | 12.2.7.4.3 | AEs: MedDRA Coding: Newborn Asian Race - Full Analysis Subject Sample | |
| AEL009 | Adverse Events | 10.1.3.1.22 | Listing of Deaths: Subject - All Subjects<br>Consented Subject Sample | |
| AEL009 | Adverse Events | 10.1.3.1.22.<br>1 | Listing of Deaths: Subject Chinese Sites - All<br>Subjects Consented Subject Sample | |
| AEL009 | Adverse Events | 10.1.3.1.22. | Listing of Deaths: Subject Asian Sites - All<br>Subjects Consented Subject Sample | |
| AEL009 | Adverse Events | 10.1.3.1.22. | Listing of Deaths: Subject Asian Race - All<br>Subjects Consented Subject Sample | |
| AEL010 | Adverse Events | 10.1.3.1.23 | Listing of Other SAEs: Subject - All Subjects<br>Consented Subject Sample | |
| AEL010 | Adverse Events | 10.1.3.1.23. | Listing of Other SAEs: Subject Chinese Sites -<br>All Subjects Consented Subject Sample | |
| AEL010 | Adverse Events | 10.1.3.1.23. | Listing of Other SAEs: Subject Asian Sites -<br>All Subjects Consented Subject Sample | |
| AEL010 | Adverse Events | 10.1.3.1.23. | Listing of Other SAEs: Subject Asian Race -<br>All Subjects Consented Subject Sample | |
| AEL010 | Adverse Events | 10.1.3.1.26 | Listing of Other SAEs: Newborn – Full<br>Analysis Subject Sample | |
| AEL011 | Adverse Events | 10.1.3.1.24 | Listing of TEAEs Leading to Study<br>Termination – Safety Subject Sample | |
| AEL011 | Adverse Events | 10.1.3.1.24. | Listing of TEAEs Leading to Study<br>Termination: Chinese Sites – Safety Subject<br>Sample | |
| AEL011 | Adverse Events | 10.1.3.1.24. | Listing of TEAEs Leading to Study<br>Termination: Asian Sites – Safety Subject<br>Sample | |

| | | | | Produced for: |
|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results |
| AEL011 | Adverse Events | 10.1.3.1.24. | Listing of TEAEs Leading to Study<br>Termination: Asian Race – Safety Subject<br>Sample | |
| AEL012 | Adverse Events | 10.1.3.1.25 | Listing of TEAEs Leading to Discontinuation of Study Drug – Safety Subject Sample | |
| AEL012 | Adverse Events | 8.3.2 | Data Portion for Subject Narratives | |
| LBL008 | Laboratory Data | 12.2.8.1 | Markedly Abnormal and/or Clinically<br>Significant Safety Laboratory Variables –<br>Safety Subject Sample | |
| LBL002 | Laboratory Data | 12.2.8.2 | Qualitative Safety Laboratory Variables - All<br>Subjects Allocated to Treatment Subject<br>Sample | |
| LBL003 | Laboratory Data | 12.2.8.3 | Quantitative Safety Laboratory Variables - All<br>Subjects Allocated to Treatment Subject<br>Sample | |
| VSL004 | Vital Signs | 12.2.8.4 | Markedly Abnormal Vital Signs – Safety<br>Subject Sample | |
| VSL005 | Vital Signs | 12.2.8.5 | Vital Signs - All Subject Allocated to<br>Treatment Subject Sample | |
| SVL001 | Subject Visits | 12.2.8.6 | Subject Visits – All Subject Allocated to Treatment Subject Sample | |
| COL001 | Comments | 12.2.9.1 | Comments – All Subjects Consented Subject<br>Sample | |

Note: A missing output code denotes a non-standard output.

## 9.2.3 Figures

For the shells of the non-standard figures, see Section 10.3.

| | | | | Produced for: |
|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline results |
| DSF001 | Subject Disposition | 10.1.4.1 | Flowchart of Subject Disposition | |
| DSF001 | Subject Disposition | 10.1.4.1.1 | Flowchart of Subject Disposition: Chinese Sites | |
| DSF001 | Subject Disposition | 10.1.4.1.2 | Flowchart of Subject Disposition: Asian Sites | |
| DSF001 | Subject Disposition | 10.1.4.1.3 | Flowchart of Subject Disposition: Asian Race | |
| DSF002 | Subject Disposition | 10.1.4.2 | Flowchart of Subject Samples | |
| EFF001 | Efficacy | 10.1.5.1 | Impact of Treatment on Pregnancy Rates – Full<br>Analysis Subject Sample | |
| EFF001 | Efficacy | 10.1.5.2 | Impact of Treatment on Pregnancy Rates – Per<br>Protocol Subject Sample | |
| EFF001 | Efficacy | 10.1.5.1a | Impact of Treatment on Pregnancy Rates by<br>Country - Full Analysis Subject Sample | |
| EFF001 | Efficacy | 10.1.5.1b | Impact of Treatment on Pregnancy Rates by<br>Age Group – Full Analysis Subject Sample | |
| EFF001 | Efficacy | 10.1.5.1c | Impact of Treatment on Pregnancy Rates by Race– Full Analysis Subject Sample | |
| EFF001 | Efficacy | 10.1.5.1d | Impact of Treatment on Pregnancy Rates by BMI – Full Analysis Subject Sample | |
| EFF001 | Efficacy | 10.1.5.1e | Impact of Treatment on Pregnancy Rates by<br>Number of Embryos transferred– Full Analysis<br>Subject Sample | |
| EFF001 | Efficacy | 10.1.5.1f | Impact of Treatment on Pregnancy Rates by<br>Weight – Full Analysis Subject Sample | |

Note: A missing output code denotes a non-standard output.